CLINICAL TRIAL: NCT02389283
Title: Sensitivity to Change of Different Reduced Ultrasound Counts in Rheumatoid Arthritis
Brief Title: Reduced Ultrasound Counts in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FIBHGM-EONC004-2014
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; ultrasound joint count
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis(RA) patients: The patients will be evaluated according to clinical practice (clinical evaluation and inflammation markers) at baseline and 3 and 6 months after the initiation of the treatment with the biologic DMARD.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease characterized by intra and peri-articular synovial inflammation. Synovitis can damage the articular cartilage, bones, joint capsule, tendons and ligaments leading to the consequential functional joint deterioration.

The main goal of RA treatment is to achieve disease remission. The treatment of RA consists of synthetic and biologic disease modifying drugs (DMARDs), being the second ones selected when low disease or remission is not achieved with the first ones. Therapeutic response monitoring in RA should be closely managed. It is classically based on clinical exploration and laboratory tests. During the last decade, the resolution improvement of musculoskeletal ultrasound (MSUS) imaging has led to the gradual incorporation of this technique in the evaluation and monitoring of patients with RA, mainly due to its better capacity to detect synovitis than clinical exploration . Ultrasound imaging is highly available, non-invasive, reproducible, affordable and well accepted by patients. Ultrasound doppler mode detects pathological synovial flow, which reflects synovial inflammation and has a demonstrated sensitivity to change in multiple longitudinal studies. Sonographic evaluation of patients with RA includes the detection of synovitis in B and Doppler mode in the joints accessible by ultrasound. There has been high variability in the literature regarding the number of joints that should be evaluated for an appropriate monitoring of the RA patients. The validity for monitoring the therapeutic response in long standing RA has been demonstrated in three reduced joint counts, including 12, 7 and 6 joints. However, in shorter evolution RA, the sensitivity to change of any of these reduced ultrasound evaluations has never been studied

DETAILED DESCRIPTION:
Primary objectives

• To evaluate the sensitivity to change of the Doppler Ultrasound evaluation of 12, 7 and 6 joints counts in RA patients with more than 6 months and less than 5 years of evolution, which initiate an effective treatment for the disease according to indication (biologic DMARD in monotherapy or combined with methotrexate).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, ≥ 18 years of age
* Patients diagnosed with RA (according to the ACR 2010 criteria) with more than 6 months and less than 5 years of active evolution and DAS28 > 3.2 or SDAI > 11, which start treatment with biologic DMARD for the first time, according to the product's summary of products characteristics (SPC).
* Patients who have granted their written informed consent for the collection and review of their data.

Exclusion Criteria:

* Patients who are already participating in a clinical trial/s at the moment of participation in this study.
* Patients with rheumatic disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients with more than 6 months and less than 5 years of active evolution (DAS28 > 3.2 or SDAI > 11) and which start treatment with biologic therapy for the first time independently of the combination with synthetic DMARDs. The patients will be evaluated according to clinical practice (clinical evaluation and inflammation markers) at baseline and 3 and 6 months after the initiation of the treatment with the biologic DMARD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Mode B and power Doppler (PD) ultrasound evaluation | at baseline and 1, 3 and 6 months after the initiation with the biologic DMARD
  Mode B and PD ultrasound evaluation will consist in quantifying the synovitis (0 to 3) in B mode (synovial hypertrophy, effusion) and PD with quantification system OMERACT (Outcome Measures in Rheumatology) in the following bilateral joints:
  * Elbows (anterior and posterior recess)
  * Carpi (radiocarpal and midcarpal + carpoulnar) (dorsal recess)
  * Second and third metacarpophalangeal (dorsal recess)
  * Second and third proximal interphalangeal of hands (dorsal and palmar recesses)
  * Knees (suprapatellar and parapatelallar recesses)
  * Tibiotalar (dorsal and lateral recesses)
  * Second and fifth metatarsophalangeal (dorsal recess)

SECONDARY OUTCOMES:
Dopler Ultrasound sensitivity to change comparison | at baseline and 1, 3 and 6 months after the initiation with the biologic DMARD

CONTACTS AND LOCATIONS:
Overall Officials: ESPERANZA NAREDO, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hopsital general Universitario Gregorio Marañón, Madrid, Madrid, Spain